CLINICAL TRIAL: NCT01597323
Title: Safety and Efficacy Evaluation of the eTWO System for Improvement of Skin Texture Via Skin Resurfacing and Wrinkles Reduction
Brief Title: Safety & Efficacy Evaluation of a Radiofrequency & Laser/Light System for Improvement of Skin Texture
Status: Completed | Type: Observational
Sponsor: Candela Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: DC84611
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Skin Texture Irregularities; Facial Skin Wrinkles
Keywords: Wrinkle Reduction; Skin Resurfacing; Skin Texture Improvement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Optional biopsy, for consenting subjects, of facial skin tissue from areas directly in front of ear (Pre-Auricular)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment Group: Healthy Male of Female between ages 35 and 60 with presence of mild to moderate facial photodamage (sun damage) and presence of mild to moderate facial wrinkling

SUMMARY:
Evaluate the clinical performance, safety and efficacy, of a Radiofrequency and Laser/Light based device for the treatment of facial wrinkles.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female between the ages of 35 and 60
2. Non-smoker
3. Fitzpatrick skin type I-VI
4. Fitzpatrick Degree of Elastosis Score of 2-6 (inclusive)
5. Presence of mild to moderate photodamage, such as solar lentigines, dyschromia and/or presence of mild to moderate facial wrinkling
6. Able and willing to comply with all visit, treatment and evaluation schedules and requirements
7. Able to understand and provide written Informed Consent
8. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment.

Exclusion Criteria:

1. Pregnant or intending to become pregnant during the course of study. A urine pregnancy test will be given to women of childbearing potential and performed during initial visit;
2. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator
3. Having a permanent implant in the treated area, such as metal plates and screws
4. Unable or unlikely to refrain from tanning, including the use of tanning booths, during the course of the study
5. Prior use of retinoids in treated area within 2 weeks of initial treatment or during the course of the study
6. Use of oral Isotretinoin (Accutane®) within 6 months of initial treatment or during the course of the study
7. Patient on systemic corticosteroid therapy 6 months prior to and throughout the course of the study
8. Having received a facial dermabrasion or chemical peel treatment within 3 months of treatment or during the study
9. Prior skin treatment with laser in treated area within 3 months of initial treatment or during the course of the study
10. Prior use of Botox, collagen, fat injections and /or other methods of skin augmentation (enhancement with injected or implanted material) in treated area within 3-4 weeks of initial treatment or during the course of the study. Treatment may not be performed at all over permanent dermal implants
11. Prior ablative resurfacing procedure, brow lift, blepharoplasty or face lift in treated area with laser or other devices within 12 months of initial treatment or during the course of the study
12. Any other surgery in treated area within 12 months of initial treatment or during the course of the study
13. History of keloid formation or poor wound healing in a previously injured skin area
14. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity)
15. Open laceration or abrasion of any sort on the area to be treated
16. Active Herpes Simplex I at the time of treatment
17. Multiple dysplastic nevi in the area to be treated
18. Having a bleeding disorder or taking anticoagulation medications, including heavy use of aspirin, in a manner which does not allow for a minimum 10 day washout period prior to the treatment (as per the subject 's physician discretion)
19. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications
20. Having any form of active cancer at the time of enrollment and during the course of the study
21. Significant concurrent illness, such as uncontrolled diabetes i.e. any disease state that in the opinion of the Investigator would interfere with the anesthesia, treatment, or healing process
22. Participation in a study of another device or drug within 1 month prior to study enrollment or during this study, and as per the Investigator's careful discretion, as long as not contradictory to any of the above criteria
23. Tattoos, including cosmetic make-up tattoos, in the treatment area
24. Mentally incompetent, prisoner or evidence of active substance or alcohol abuse
25. Any condition which, in the Investigator's opinion, would make it unsafe (for the subject or for the study personnel) to treat the subject as part of this research

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Male of Female between ages 35 and 60 with presence of mild to moderate facial photodamage (sun damage) and presence of mild to moderate facial wrinkling
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2011-10-25 (Actual); Primary Completion 2014-10-14 (Actual); Study Completion 2014-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan H Gold, MD, Principal Investigator — Board Certified Plastic Surgeon, American Board of Plastic Surgeons; Robert Weiss, MD, Principal Investigator — Board Certified Dermatologist, American Board of Medical Specialties; Jason N Pozner, MD, Principal Investigator — Board Certified Plastic Surgeon, American Board of Plastic Surgeons
Locations (3):
- United States (3):
  - Sanctuary Medical Aesthetic Center, Boca Raton, Florida
  - The Maryland Laser, Skin and Vein Institute, Hunt Valley, Maryland
  - Cosmetic & Reconstructive Plastic Surgery, Great Neck, New York